CLINICAL TRIAL: NCT07396064
Title: Bridging the Gap: Enhancing Cancer Care for Underserved Populations With the Veris Health Cancer Care Platform
Status: Not yet recruiting | Type: Observational
Sponsor: VERIS HEALTH INC (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Organization: PAVmed Inc. (Industry)
Other Study IDs: VER-PR-0023; 5R44MD019611-02 (NIH)
Record Dates: First submitted 2026-01-27; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Cancer Care Recipient; Observational Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main Phase group: All participating subject utilizing the Veris Health app will complete all study health measurements with a 24 week period on the Veris Health app as well as participate in interviews and focus groups.
  Interventions: Other: Veris Health Inc. Application

INTERVENTIONS:
Other: Veris Health Inc. Application — Veris Health offers at-home devices to monitor multiple physiological parameters, including temperature, heart rate, oxygen saturation, blood pressure, weight, and activity (step count). Patients are provided with a home cellular hub that is already paired to peripheral devices via Bluetooth. The hub communicates with all devices and the local cellular network out-of-the-box, and data is automatically sent via cellular network to the Veris Health backend database, making it easy for patients to use the system. Patients are responsible for taking their vital sign measurements daily. The devices automatically send the measurement data to the Veris Health HIPAA compliant, secure cloud server via the preconnected cellular hub.

SUMMARY:
The proposed study aims to optimize and validate the Veris Cancer Care Platform for the needs of medically underserved cancer patients receiving outpatient cancer therapy. The Veris Health platform is a remote patient monitoring and communication system designed to bridge the gap between clinical visits and provide oncology care teams with objective data during high-risk periods.

This study will specifically focus on optimizing the Veris Health platform for patients with language barriers, limited access to technology, and socioeconomic disparities. By incorporating user-centered design and working closely with community health centers, the research team will ensure that the platform is culturally and linguistically appropriate, easy to use, and accessible for all patients.

The study will use a mixed-methods approach to validate the effectiveness of the optimized platform, including quantitative data analysis and qualitative interviews with patients and healthcare providers. The goal is to demonstrate the potential for the Veris Health platform to improve outcomes for vulnerable populations by reducing hospitalizations, emergency department visits, and the economic burden of cancer care.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years old
* Diagnosis of cancer
* ECOG Performance Status of 0-2
* Undergoing or initiating systemic anticancer therapy
* Able to utilize and interact with a mobile application and in-home devices for physiological monitoring. Have at least one of the following barriers to healthcare access: Spanish as primary language, uninsured, insured with Medicaid, dual eligible for Medicare and Medicaid

Exclusion Criteria:

-N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Underserved population undergoing Cancer treatment with at least one on the following barriers to healthcare access: Spanish as primary language, uninsured, insured with Medicaid, dual eligible for Medicare and Medicaid.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Usability of the Veris Health Cancer Care Platform | 5 Months
  Usability of the Veris Health Cancer Care platform as assessed by the Software Usability Measurement Inventory (SUMI) among patients, caretakers, and healthcare teams.
  Measure: SUMI total and domain scores
  Time Frame: During study participation
Product Design Usability and Acceptability | 5 Months
  Ease of use, accessibility, and acceptability of the Veris Health Cancer Care platform based on A/B testing of product design features.
  Measure: Comparative usability metrics (e.g., task completion success, user preference)
  Time Frame: During study participation
User Needs and Preferences | 5 Months
  User-identified needs, preferences, and barriers to use of the Veris Health Cancer Care platform.
  Measure: Qualitative themes derived from user interviews and focus groups
  Time Frame: During study participation

SECONDARY OUTCOMES:
Health-Related Quality of Life (HRQL) | 5 Months
  Change in health-related quality of life among participants using the Veris Health Cancer Care platform.
  Measure: EQ-5D Index score
Symptom Burden of Cancer Treatment Side Effects | 5 Months
  Frequency and severity of cancer treatment-related symptoms, including nausea, diarrhea, and infection.
  Measure: Patient-reported symptom frequency and severity scores
Cancer Treatment Adherence and Duration | 5 months
  Adherence to prescribed cancer therapy and treatment duration.
  Measure: Rates of dose reductions, early treatment discontinuation, and treatment duration

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.verishealth.com